CLINICAL TRIAL: NCT04075903
Title: Improving Care for Gout in the Southeast Enhancing Gout Minority Patients Care and Participation in Gout Clinical Research
Brief Title: Gout in the ED and Improving Research Participation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Massachusetts General Hospital (Other); MetroHealth Medical Center (Other); University of Iowa (Other); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Kenneth Saag, MD, MSc, Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 300003869; P50AR060772 (NIH)
Record Dates: First submitted 2019-08-29; First posted 2019-09-03 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Storytelling A health literacy-appropriate and culturally-adapted intervention delivered on a tablet computer containing "storytelling" to improve patient gout knowledge and approaches to prevent flares, destigmatize gout, and enhance readiness to adopt available long-term treatments for gout including medications, diet, and exercise, or ii) usual gout care (control state).
  Interventions: Behavioral: Storytelling
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Storytelling — A health literacy-appropriate and culturally-adapted intervention delivered on a tablet computer containing "storytelling" to improve patient gout knowledge and approaches to prevent flares, destigmatize gout, and enhance readiness to adopt available long-term treatments for gout including medications, diet, and exercise, or ii) usual gout care (control state).
  Arms: Intervention

SUMMARY:
The prevalence of gout has been steadily increasing over several decades and is correlated with the rising burden of obesity, chronic cardiac and renal disease; all conditions overrepresented in the Southeastern U.S. - particularly in African Americans. Through a novel emergency department led intervention we aim to improve the care patients with gout receive, both during acute exacerbations and long-term. A secondary goal of the project is to concurrently enhance participation of minorities in biomedical research in the Deep South.

DETAILED DESCRIPTION:
Gout is a chronic disease that affects over 9 million Americans. It is characterized by intermittent flares associated with severe pain. The prevalence of gout has been steadily increasing over several decades and it correlates with the rising burden of obesity, chronic cardiac and renal disease, all conditions overrepresented in the Southeastern U.S. - particularly in African Americans. In addition, many gout patients are not adherent with their follow-up visits due to a lack of awareness of the consequences of untreated gout and/or poor access to health care. As a result, US emergency departments (EDs) are delivering an increasing amount of gout care for underserved populations.

To address this significant public health problems teams at the University of Alabama at Birmingham (UAB), University of Iowa, Massachusetts General Hospital (MGH), and MetroHealth Medical Center are collaborating on a novel emergency department-led intervention aimed at improving the gout care patients receive, during periods of acute flare and long-term. Investigators hypothesize that the use of educational material including cultural appropriate stories about what it is like to live with gout and the use of navigators who will help patients better coordinate their care, will be associated with improved rates of patients that have a follow-up visit addressing gout after the ED visit. A secondary goal is to enhance participation of underrepresented minorities in biomedical research in the Deep South as part of an NIH funded gout center at UAB.

Investigators will recruit and enroll adults (at least 18 years of age) that have confirmed gout. Participants will include men and women of all races/ethnicities. Recruitment will occur in the EDs at UAB, University of Iowa, MGH, and MetroHealth. Qualifying patients will be assigned by chance to get either 1) our enhanced educational materials coupled (at UAB) with a lay person who can help them coordinate their care or 2) to receive the current usual standard of care for their gout. After a gout diagnosis is confirmed by a research assistant, informed consent will be obtained. Following enrollment, participants will complete questionnaires at 3 and 6 months. Beyond follow-up visits, Investigators will also measure differences in the groups between the use of medication for gout treatment, other healthcare visits, changes in weight, satisfaction, and overall health during study follow-up. Leveraging the resources of UAB, including the National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) funded Center of Research Translation (CORT) in gout and hyperuricemia and ongoing collaborations between these medical institutions, Investigators have assembled a multidisciplinary scientific team, uniquely prepared to execute the proposed study to help medically underserved gout patients and enhance research diversity in the Southeast.

ELIGIBILITY:
Inclusion Criteria:

* Gout diagnosis meeting 2015 American College of Rheumatology and European League Against Rheumatism classification criteria,99,140
* Adult > 18 years of age
* Able to communicate and understand English language (a future objective, with additional resources, will include Spanish translation of all study materials).

Key exclusion criteria:

* Joint complaint related to significant trauma or recent surgery (<1 month)
* Life expectancy of < 6 months
* Current critical illness leading to admission to high acuity medical care unit (ICU, stepdown unit) or requiring surgical intervention (general anesthesia); confirmed septic arthritis or joint infectious arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2026-02-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - MetroHealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
We are prepared to share data in the following ways: (a) perform a final data edit on the complete data set; (b) create a final data file; (c) perform statistical analyses that support the study findings; (c) issue final reports to the appropriate authorities and collaborators; and (e) provide copies of the finalized data sets. The finalized datasets will be made public with the requisite documentation. All datasets made public will be distributed first to all collaborating co-investigators for verification and testing. The mode of dissemination of these public datasets will be via archive files accessible in the public domain. Public datasets will be de-identified so that they are free of all identifiers that would permit linkages to individual research participants and of variables that could lead to deductive disclosure of the identity of individual participants. Bio-specimens collected and stored as part of this study will be made available through requests to the INSIGHT CORT.

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Storytelling and Navigation A health literacy-appropriate and culturally-adapted intervention delivered on a tablet computer containing "storytelling" to improve patient gout knowledge and approaches to prevent flares, destigmatize gout, and enhance readiness to adopt available long-term treatments for gout including medications, diet, and exercise, along with post-emergency department visit patient navigation to promote outpatient follow-up
Period: Overall Study
Arm/Group | Intervention | Control
Started | 135 | 65
Completed | 135 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 135 | 65 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (13.6) | 58.9 (12.4) | 58 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 15 | 49
  Male | 101 | 50 | 151
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 92 | 45 | 137
  White | 35 | 16 | 51
  Asian, Hispanic or Latino, Unknown/Other | 8 | 4 | 12
Education Level [Count of Participants; unit: Participants]
  High School Graduate or Less | 65 | 30 | 95
  Vocational Training or Some College | 44 | 23 | 67
  4-year Degree or More Completed | 23 | 12 | 35
Employment Status [Count of Participants; unit: Participants]
  Full-Time Work | 61 | 19 | 80
  Part-Time Work or Not Seeking Work | 37 | 22 | 59
  Unemployed | 25 | 16 | 41
  Other or Choose not to Answer | 8 | 8 | 16
Yearly Income [Count of Participants; unit: Participants]
  Less than $30,000 | 42 | 20 | 62
  $30,000 to less than $60,000 | 13 | 13 | 26
  $60,000 to less than $100,000 | 14 | 8 | 22
  Greater than $100,000 | 11 | 4 | 15
  Prefer not to answer | 44 | 18 | 62
Smoking Status [Count of Participants; unit: Participants]
  Currently Smoking Everyday | 17 | 9 | 26
  Currently Smoking Some Days | 18 | 4 | 22
  Not Smoking at All | 97 | 50 | 147
Alcohol Use [Count of Participants; unit: Participants]
  2 or more times per week | 24 | 10 | 34
  2-4 times per month | 53 | 22 | 75
  Never | 54 | 33 | 87

OUTCOME MEASURES:

1. Primary Outcome: Outpatient Primary Care or Specialist Visits for Gout Treatment
Description: Proportion of participants who attend a primary care or specialist visits for gout treatment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 135 | 65
Participants
  Presence of Gout Follow-Up | 64 | 35

ADVERSE EVENTS:
Time Frame: 3 months
Description: This was a minimal risk study. No adverse events or serious adverse events were reported during follow-up outcomes assessment.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/65
Other Adverse Events (participants affected / at risk) | 0/135 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT04075903/Prot_SAP_000.pdf